CLINICAL TRIAL: NCT05822167
Title: Effect of Food Temperature and Diet Composition on Satiety, Satiety Hormones, Chewing Time and Neuronal Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Bibi Hajira, Assistant Professor, Khyber Medical University Peshawar
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KMU/IBMS/IERB/2022/9303-7
Record Dates: First submitted 2023-03-06; First posted 2023-04-20 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Obesity, Overweight
Keywords: Satiety; Food Intake; Food Temperature; Food Composition; Gut Hormones; Satiety-related Hormones; Chewing time; Appetite; Satiety Score; EEG; Brain Waves; EMG; CCK; GLP-1; Insulin; Peptide YY; Ghrelin; high Protein meal; high Fat meal; High Carbohydrate meal; Chewing count; Alpha wave
MeSH Terms: conditions — Obesity; Overweight; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: 3 interventional Studies 9 arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- High Protein Meal with cold temperature (Experimental)
  Interventions: Other: High Protein Meal at Cold Temperature
- High Protein Meal with warm temperature (Experimental)
  Interventions: Other: High Protein Meal at Warm Temperarute
- High Protein Meal with Hot temperature (Experimental)
  Interventions: Other: High Protein Meal at Hot Temperature
- High Carbohydrate Meal with cold temperature (Experimental)
  Interventions: Other: High Carbohydrate Meal at Cold Temperature
- High Carbohydrate Meal with warm temperature (Experimental)
  Interventions: Other: High Carbohydrate Meal at Warm Temperature
- High Carbohydrate Meal with hot temperature (Experimental)
  Interventions: Other: High Carbohydrate Meal at Hot Temperature
- High Fat Meal with cold temperature (Experimental)
  Interventions: Other: High Fat Meal at Cold Temperature
- High Fat Meal with warm temperature (Experimental)
  Interventions: Other: High Fat Meal at Warm Temperature
- High Fat Meal with hot temperature (Experimental)
  Interventions: Other: High Fat Meal at Hot Temperature

INTERVENTIONS:
Other: High Protein Meal at Cold Temperature — High Protein Meal providing 500kcal with 60% energy from protein, 30% fat, 10% carbohydrate.
  Cold meal will be served at 25 degree C and below.
  Arms: High Protein Meal with cold temperature
Other: High Protein Meal at Warm Temperarute — High Protein Meal providing 500kcal with 60% energy from protein, 30% fat, 10% carbohydrate.
  Meal will be served at warm temperature i.e., between 40 degree C and 60 degree C.
  Arms: High Protein Meal with warm temperature
Other: High Protein Meal at Hot Temperature — High Protein Meal providing 500kcal with 60% energy from protein, 30% fat, 10% carbohydrate.
  Meal will be served at hot temperature i.e., 60 degree C and above.
  Arms: High Protein Meal with Hot temperature
Other: High Carbohydrate Meal at Cold Temperature — High carbohydrate meal providing 500 kcal with 65% of energy from carbohydrates, 25% from proteins and 10% from fats.
  Cold meal will be served at 25 degree C and below.
  Arms: High Carbohydrate Meal with cold temperature
Other: High Carbohydrate Meal at Warm Temperature — High carbohydrate meal providing 500 kcal with 65% of energy from carbohydrates, 25% from proteins and 10% from fats.
  Meal will be served at warm temperature i.e., between 40 degree C and 60 degree C.
  Arms: High Carbohydrate Meal with warm temperature
Other: High Carbohydrate Meal at Hot Temperature — High carbohydrate meal providing 500 kcal with 65% of energy from carbohydrates, 25% from proteins and 10% from fats.
  Meal will be served at hot temperature i.e., 60 degree C and above.
  Arms: High Carbohydrate Meal with hot temperature
Other: High Fat Meal at Cold Temperature — High fat meal will contain 60% fat, 30% protein, 10% carbohydrate. Cold meal will be served at 25 degree C and below.
  Arms: High Fat Meal with cold temperature
Other: High Fat Meal at Warm Temperature — High fat meal will contain 60% fat, 30% protein, 10% carbohydrate. Meal will be served at warm temperature i.e., between 40 degree C and 60 degree C.
  Arms: High Fat Meal with warm temperature
Other: High Fat Meal at Hot Temperature — High fat meal will contain 60% fat, 30% protein, 10% carbohydrate. Meal will be served at hot temperature i.e., 60 degree C and above.
  Arms: High Fat Meal with hot temperature

SUMMARY:
Obesity and its related illnesses have become serious health issues, obesity is today the fifth most common cause of death. Obesity rate has dramatically enhanced in both male and female, and across all ages. Food and energy intake during habitual meals, energy balance, energy expended during physical activity, all play an important role in management of weight.

Lifestyle changes and nutritional strategies are emerging as the best line of treatment for obesity. The achievement of satiety along with, the reduction in dietary intake is the primary goal of nutritionists and food scientists. Appetite control can be defined by two terms; satiety and satiation. The interaction between appetite, food intake, and hormones secreted by the gastrointestinal tract, which are secreted in response to macronutrients like carbohydrates, fats and proteins are the satiety regulators. The gut hormones including glucagon like peptide 1(GLP1), cholecystokinin (CCK) are anorexigenic in action, cause slowing of meal digestion and reduce food intake thus inducing satiation and satiety. The CCK hormone plays a key role in delaying of stomach emptying by fundus relaxation and antral inhibition, ultimately causing major satiation. The incretin hormone GLP-1's main action is to stimulate insulin secretion, inhibit glucagon secretion, regulating postprandial glucose and provide negative feedback to the stomach thereby controlling appetite. Research is needed in meal properties and different diets which may affect gut-brain signaling and altering the mechanisms of gut hormonal secretion, thus further influencing appetite satiation and satiety scores. This knowledge can be utilized in energy expenditure and weight management.

Serving temperatures alter perceived intensities, flavor and acceptances of food as well. Brain areas work in close association with the thermal perception and emotions. In neuroimaging studies neural changes have been when body is exposed to different temperatures either environmental or oral cavity. Temperature of food play an important role in the palatability and affective value of food and, consequently, in appetite regulation. Limited research has been done so far how food temperature is related to sensory perception and satiety Chewing and food texture also affect satiety and satiation. The oral processing, eating rate and physical forms of food i.e., solid versus liquid or semi-solid are all physiologically related to satiety and an individual's behavior to understand this oral sensory satiety effect, requires further studies. The number of chews has been studied showing an association between reduction in food intake with increasing number of chews. EEG is a noninvasive neuroimaging technique, helping in evaluating the cognitive part of food stimuli and food ingestion in relation to gut hormones. Sensory properties of previously identified as drivers of refreshing perception, enhance alpha and beta brain oscillations as observed in prior EEG studies.

Many factors influence satiety including food composition, temperature, environment, last meal and preload. Limited literature is available about temperature of food and its influence on satiety. My study aims to find 1) the effect of temperature of high carbohydrate, high fat meal and high protein meal on the satiety scores, satiety-related hormones, EEG and EMG. 2. To find the effect of chewing time of food on the satiety scores, satiety- related hormones, EEG and EMG.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals of age 25- 35 years
* BMI ranged between 18.5 and 24.9

Exclusion Criteria:

* Chronic diseases, diabetes, endocrine disorder,
* Any bariatric surgery that interfered with gastrointestinal functions,
* Smoking,
* Dieting,
* Pregnancy, lactation,
* Taking medication or supplements.
* Psychiatry illnesses or dental problems will be excluded.
* Females with the history of premenstrual syndrome will be excluded.
* Gastrointestinal Complications
* Following Special diets
* Food allergy to food used in the trial

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Hedonic 9-point | 30 minutes
  Hedonic 9-point scale for acceptability of meal in terms of appearance, texture, smell, flavor and temperate.
GLP-1 | Change from baseline till 4 hours
  Glucagon like peptide-1
Chew Counting | Up to 2 hours
  Chew Counting was done while the test meal is consumed by the participant by EMG and video recording same time.
EEG | Change from baseline till 1 hour
  Pre-prandial baseline EEG was done and then immediately after when the food intake is finished and 1 hour post prandial. Alpha wave amplitude and frequency were noted.
CCK | 0 minutes, 30 minutes and 180 minutes
  Cholecystokinin
PYY | Change from baseline to 180 minutes
  Peptide tyrosine tyrosine
Ghrelin | Change from baseline to 120 minutes
  Human ghrelin
Glucose | Change from baseline to 120 minutes
  Pre-prandial baseline glucose and then after food intake
Insulin | Change from baseline to 180 minutes
  Pre-prandial baseline and after food intake
Serotonin | Change from baseline to 60 minutes
  Pre-prandial baseline and after food intake

SECONDARY OUTCOMES:
Remainder food intake | Up to 24 hours
  The food given to the subjects was weighed before serving. After the participants had finished their meals the serving dish with the left overs was weighed again with the kitchen weighing scale.
Satiety | Change from baseline to 240 minutes
  Visual analog scale on a scale of 0 to 100 mm. High score indicate better and low score indicate worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Medical University, Peshawar, KPK, Pakistan

REFERENCES:
- [Background] Rexrode KM, Carey VJ, Hennekens CH, Walters EE, Colditz GA, Stampfer MJ, Willett WC, Manson JE. Abdominal adiposity and coronary heart disease in women. JAMA. 1998 Dec 2;280(21):1843-8. doi: 10.1001/jama.280.21.1843. PMID 9846779
- [Background] McMillan DC, Sattar N, McArdle CS. ABC of obesity. Obesity and cancer. BMJ. 2006 Nov 25;333(7578):1109-11. doi: 10.1136/bmj.39042.565035.BE1. No abstract available. PMID 17124223
- [Background] Chambers L, Mc Crickerd K, Yeomans M. R. Optimising foods for satiety.Trends Food Sci. Technol. 2015; 41: 149-160. https ://doi.org/10.1016/j.tifs.2014.10.007
- [Background] Blundell J. E, De Graaf K , Finlayson G, Halford J. C, Hetherington M, KingN, & Stubbs J. Assessment Methods for Eating Behaviour and Weight-Related Problems: Measures, Theory and Research. 2009; 283-325 (Sage, Thousand Oaks).
- [Background] Camilleri M. Peripheral mechanisms in appetite regulation. Gastroenterology. 2015 May;148(6):1219-33. doi: 10.1053/j.gastro.2014.09.016. Epub 2014 Sep 21. PMID 25241326
- [Background] van der Klaauw AA, Keogh JM, Henning E, Trowse VM, Dhillo WS, Ghatei MA, Farooqi IS. High protein intake stimulates postprandial GLP1 and PYY release. Obesity (Silver Spring). 2013 Aug;21(8):1602-7. doi: 10.1002/oby.20154. Epub 2013 May 13. PMID 23666746
- [Background] Strader AD, Woods SC. Gastrointestinal hormones and food intake. Gastroenterology. 2005 Jan;128(1):175-91. doi: 10.1053/j.gastro.2004.10.043. PMID 15633135
- [Background] Gibbons C, Finlayson G, Caudwell P, Webb DL, Hellstrom PM, Naslund E, Blundell JE. Postprandial profiles of CCK after high fat and high carbohydrate meals and the relationship to satiety in humans. Peptides. 2016 Mar;77:3-8. doi: 10.1016/j.peptides.2015.09.010. Epub 2015 Sep 30. PMID 26429068
- [Background] Tanaka M, Nagashima K, McAllen RM, Kanosue K. Role of the medullary raphe in thermoregulatory vasomotor control in rats. J Physiol. 2002 Apr 15;540(Pt 2):657-64. doi: 10.1113/jphysiol.2001.012989. PMID 11956351
- [Background] Rolls ET. The affective and cognitive processing of touch, oral texture, and temperature in the brain. Neurosci Biobehav Rev. 2010 Feb;34(2):237-45. doi: 10.1016/j.neubiorev.2008.03.010. Epub 2008 Apr 3. PMID 18468687
- [Background] Miquel-Kergoat S, Azais-Braesco V, Burton-Freeman B, Hetherington MM. Effects of chewing on appetite, food intake and gut hormones: A systematic review and meta-analysis. Physiol Behav. 2015 Nov 1;151:88-96. doi: 10.1016/j.physbeh.2015.07.017. Epub 2015 Jul 15. PMID 26188140
- [Background] Robinson E, Almiron-Roig E, Rutters F, de Graaf C, Forde CG, Tudur Smith C, Nolan SJ, Jebb SA. A systematic review and meta-analysis examining the effect of eating rate on energy intake and hunger. Am J Clin Nutr. 2014 Jul;100(1):123-51. doi: 10.3945/ajcn.113.081745. Epub 2014 May 21. PMID 24847856
- [Background] Schlogl H, Horstmann A, Villringer A, Stumvoll M. Functional neuroimaging in obesity and the potential for development of novel treatments. Lancet Diabetes Endocrinol. 2016 Aug;4(8):695-705. doi: 10.1016/S2213-8587(15)00475-1. Epub 2016 Jan 30. PMID 26838265
- [Background] Hallschmid M, Molle M, Fischer S, Born J. EEG synchronization upon reward in man. Clin Neurophysiol. 2002 Jul;113(7):1059-65. doi: 10.1016/s1388-2457(02)00142-6. PMID 12088700